CLINICAL TRIAL: NCT06808035
Title: Understanding Perinatal Spinal Cord Injury: Comprehensive Assessment and Personalized Neuromodulation for Improved Whole-Body Functions
Brief Title: Understanding Perinatal Spinal Cord Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Vanderbilt University (Other); University of Leeds (Other); Kentucky Spinal Cord and Head Injury Research Trust (Unknown)
Responsible Party: Principal Investigator, Andrea L. Behrman, PhD, PT, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23.0722
Record Dates: First submitted 2024-12-12; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Perinatal Spinal Cord Injury
Keywords: Spinal Cord Injury; Activity-Based Recovery Training; Perinatal-Onset; Transcutaneous Spinal Cord Stimulation; Whole-Systems; Pediatric Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cervical Perinatal SCI (Experimental): Participants with high cervical and low cervical SCI will perform tailored ABRT+scTS. Pre, interim, and post assessments of neurophysiological, sensorimotor, and autonomic function will be compared within-subjects and between high and low cervical SCI groups. Participants will come for daily activity-based recovery training (ABRT) + transcutaneous spinal stimulation (scTS). ABRT+scTS will take place 5 days per week for approximately 2.5 hours each (1.5 hours of lower extremity training and 1 hour of upper extremity training) for a total of 40 sessions consisting of facilitated sitting, standing, stepping, and UE motor tasks such as grasping, reaching, and hand manipulations.
  Interventions: Other: Activity-Based Recovery Training; Device: Transcutaneous Spinal Cord Stimulation

INTERVENTIONS:
Other: Activity-Based Recovery Training — ABRT uses task-specific training to improve neuromuscular capacity. ABRT will be tailored to participant presentation. Activity-Based Locomotor Training consists of stepping, standing, and sitting activities on a body weight support (BWS) treadmill using a harness and while overground. Therapists and trainers provide hands-on assistance for safety and kinematics. BWS is varied during sessions with a goal of optimal kinematics at the lowest BWS. Activities performed standing will focus on alignment incorporating static, active, and dynamic tasks. Activities performed during overground are based on neuromuscular capacity and appropriate developmental and functional levels. Principles of ABRT will be shared with parents/caregivers to foster activity in the home and community. Activity-Based Upper Extremity Training uses task-specific training of the trunk and upper extremities administered in sitting or standing via manual facilitation or support in a stander for best posture.
  Other Names: Activity-Based Training; Activity-Based Locomotor Training; Activity-Based Upper Extremity Training; ABRT; ABT; AB-LT; AB-UET
Device: Transcutaneous Spinal Cord Stimulation — Transcutaneous Spinal Cord Stimulation (scTs) is a non-invasive stimulation administered over the skin using a modulated biphasic or monophasic waveform at 15-90Hz and a carrier frequency of 5-10kHz. Bouts of scTs at the cervical, thoracic, lumbar, and/or coccygeal level will be administered midline or just lateral to the spinous processes during activity-based recovery training.
  Other Names: scTS; TcStim

SUMMARY:
The purpose of this study is to deepen our understanding of children who have a cervical spinal cord injury obtained in utero or at birth and examine the effects of tailored activity-based recovery training (ABRT) in combination with transcutaneous spinal cord stimulation (scTS). This is a within subjects, pre-post design study. Neurophysiological, sensorimotor, and autonomic assessments will occur pre, interim, and post 40 sessions of ABRT in conjunction with scTs.

DETAILED DESCRIPTION:
Infants who suffer perinatal spinal cord injuries (SCI) are injured during a critical period of neurological development. Confounded further by on-going development, they are particularly vulnerable to the consequences of SCI (e.g., paralysis and paresis, hypertonia, bladder/bowel dysfunction, respiratory compromise) on lifelong health, function, and quality of life. There are only 4 published case reports of the presentation and rehabilitation of perinatally injured children. Clinically, children with high cervical SCI compared to those with low level SCI exhibit slow and limited active upper and lower extremity (UE, LE) movements, high tone, and poor trunk control. Children with low cervical lesions have a more typical pattern of loss below the injury level. We intend to expand our understanding of the scope of perinatal SCI and its impact in order to address integrated, whole-body system rehabilitation.

The overall objective of this study is to deepen our understanding of pediatric perinatal cervical SCIs and then formulate tailored treatment strategies that encourage neuroplasticity, enhance functional capacity, and improve the overall quality of life of children. The results from this study will provide pilot data and evidence that we can comprehensively assess and develop a therapeutic roadmap to improve whole-body function in children with perinatal SCI.

This is a pilot, within subjects, repeated measures, pre-post design.

Aim 1: Investigate the impact of perinatal, cervical SCI comparing high (C2-3) and low (C4-6) injuries on a whole-body profile of health: neurophysiological, sensorimotor, autonomic.

Aim 2: In children with perinatal SCIs, investigate the effect of 40 sessions of tailored transcutaneous spinal stimulation (scTS) paired with activity-based restorative therapies (ABRTs) on neurophysiological profile (spinal pathway functional integrity) and sensorimotor function.

Aim 3: In children with chronic, cervical, perinatal SCIs, investigate the effect of 40 sessions of scTS paired with ABRT on autonomic functions, i.e., respiratory, blood pressure regulation, bladder/bowel.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with a perinatal (injured in utero or at birth), upper motor neuron spinal cord injury involving cervical spinal levels
* discharged from inpatient hospitalization/inpatient rehabilitation

Exclusion Criteria:

* Botox use within the past 3 months
* Current oral baclofen or baclofen pump use
* Musculoskeletal impairment limiting range of motion (e.g. severe scoliosis), unhealed fracture, or other medical impairment limiting study participation
* History of allodynia (heightened skin sensitivity typically at the level of the lesion site)
* History of scoliosis surgery
* Ventilator-dependence
* Unwillingness to wean from daytime use of thoroco/lumbosacral orthosis and ankle/foot orthosis during the intervention period

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Participant Specific Outcome Measures | At study enrollment, following 20 sessions (approximately 1 month), and following 40 sessions (approximately 2 months)
  Participant specific outcomes measures will be identified at study initiation via parent interview. Parents will identify daily, functional tasks that the participant has difficulty or challenges performing at a practical, successful level. Functional tasks performed by the participant will be video recorded at study initiation, post-20 sessions, and post-40 intervention sessions. Metrics of task performance include success or failure of the task.

SECONDARY OUTCOMES:
Supine Functional Neurophysiological Assessment (FNPA) | At study enrollment and following 40 sessions (approximately 2 months)
  1) Averaged electromyography (EMG) root mean square (RMS) values above and below the level of the lesion. 2) EMG isolated to limb performing the task and proximal stabilizers (yes, no). If no, identify location (limbs/trunk) of auxiliary EMG activity, 3) Timing of response
Acoustic Startle Response (ASR) | At study enrollment and following 40 sessions (approximately 2 months)
  Percent of responses above (blink) and below the level of the lesion.
Somatosensory Evoked Potentials (SSEP) | At study enrollment and following 40 sessions (approximately 2 months)
  1. Presence of response in the brain from stimulation of tibial and median nerves in the periphery, below and above the spinal cord lesion.
  2. If response is present, latency of responses (mseconds) from initiation of stimulation and across the lesion.
Stand/Step Functional Neurophysiological Assessment (FNPA) | At study enrollment and following 40 sessions (approximately 2 months)
  Test completed in children who are non-ambulatory.
  1) Can child initiate a step in the treadmill environment with body weight support? From parallel stance: Yes or No. From stride stance: Yes or No. if yes, hip range of motion (degrees) during swing.
Upper Extremity Motor Control Assessment | At study enrollment and following 40 sessions (approximately 2 months)
  Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) scores, Box and Block Test (BBT( number of blocks), transer BBT time (tBBT), hand grip force, pinch force
Trunk Motor Control Assessment | At study enrollment and following 40 sessions (approximately 2 months)
  Averaged electromyography RMS values of the trunk muscles, trunk posture (angles)
Segmental Assessment of Trunk Control | At study enrollment, following 20 sessions (approximately 1 month), and following 40 sessions (approximately 2 months)
  Score between 1-20 indicating the level of appropriate static, active, and reactive control of the trunk and level of support described.
Pediatric Neuromuscular Recovery Scale (NRS) | At study enrollment, following 20 sessions (approximately 1 month), and following 40 sessions (approximately 2 months)
  Overall and individual task NRS scores. Units of 1A-4C
Spasticity of upper extremity and lower extremity | At study enrollment, following 20 sessions (approximately 1 month), and following 40 sessions (approximately 2 months)
  Number of cycles elicited in response to the pendulum drop-test
Respiratory Motor Control Assessment (RMCA) | At study enrollment and following 40 sessions (approximately 2 months)
  Lung volume, maximum inspiratory pressure, maximum expiratory pressure, and peak cough flow will be reported.
Bowel Questionnaire | At study enrollment and following 40 sessions (approximately 2 months)
  Total Neurogenic Bowel Dysfunction (NBD) score and interpretation of impairment: 0-6 Very Minor, 7-9 Minor, 10-13 Moderate, 14+ Severe neurogenic bowel dysfunction.
Overground Walking Assessment of Gait | At study enrollment and following 40 sessions (approximately 2 months)
  1. Observational Gait Scale (OGS) Tool - score out of 22
  2. Spinal Cord Injury Functional Ambulation Inventory (SCI-FAI) Category Scores
Bladder Questionnaire | At study enrollment and following 40 sessions (approximately 2 months)
  A change in lower urinary tract function within the study timeframe per variable from an impaired state to recovery will be reported, specifically: Awareness of need to empty the bladder, bladder emptying methods, average number of voluntary bladder emptying, involuntary urine leakage, a change in medication, surgical procedures.
Gross Motor Function Measure-88 (GMFM-88) | At study enrollment and following 40 sessions (approximately 2 months)
  88 tasks across 5 dimensions: 1. lying/rolling, 2) sitting, 3) crawling/kneeling, 4) standing, 5) walking/running/jumping. Individual item scores (0-3, not tested (NT), dimension percentage, and overall percentage will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD of demographics and primary and secondary outcomes measures will be shared via Open Data Commons for Spinal Cord Injury.
Time Frame: IPD will be made available beginning 1 year after publication with no end date.
Access Criteria: Authorized users who have acquired an OCD account will have access to IPD.
URL: https://odc-sci.org/

REFERENCES:
- See also: Related Info — https://victoryoverparalysis.org/